CLINICAL TRIAL: NCT01985919
Title: Protocol for Facilitating the Acquisition of Research Bone Marrow and Blood Samples
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 01709
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: No Restrictions on Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone marrow aspirate/biopsy and blood specimens: Collection of blood and bone marrow specimens for research purposes and increase the successful acquisition of correlative bone marrow samples to improve translational research in bone marrow diseases
  Interventions: Other: Obtaining human tissue for basic research or biospecimen bank

INTERVENTIONS:
Other: Obtaining human tissue for basic research or biospecimen bank

SUMMARY:
This clinical research protocol is intended to allow for bone marrow aspirate/biopsy and blood specimens to be collected for research purposes, specifically allowing subjects the option of sedation during the bone marrow procedure. Samples will be banked for future research related to cancer and other diseases. Researchers hope this protocol will improve the collection of research correlative and translational biopsy specimens for clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Planned procedure including a bone marrow aspirate and/or bone marrow biopsy
* The procedure is planned for the purpose of obtaining a research specimen (as part of another research study or as part of this stand-alone sample collection protocol.). Procedures with a dual purpose (i.e. to obtain both clinically-indicated specimens and research specimens) are permitted, but procedures to obtain clinical specimens only are not permitted.
* All subjects must provide written informed consent for the biopsy procedure, the collection of bone marrow and blood specimens for research purposes and (if planned) the administration of sedation.

Exclusion Criteria:

* Moderate sedation may not be administrated to subjects with a clinical contraindication to its provision, or if the investigator believes that administration of moderate sedation would constitute under risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and females, 18 years of age and older who are scheduled to undergo a bone marrow aspirate and/or bone marrow biopsy as part of their participation on another research study, who are allowing their samples to be collected and used for research purposes, and/or who might benefit from the administration of moderate sedation. Therefore, there are no restrictions with regards to diagnosis, though most patients will have hematologic malignancies (leukemia, lymphoma, myeloma, amyloidosis, myelodysplastic syndromes, myeloproliferative diseases).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-02-01 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dan Vogl, MD, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States